CLINICAL TRIAL: NCT03860779
Title: Biopotentials for Clinician Satisfaction With Sedation in Colonoscopy
Acronym: BCSSC
Status: Completed | Type: Observational
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Alexander Hann, Senior Gastroenterologist, Department of Gastroenterology, University of Ulm
Other Study IDs: BCSSC
Record Dates: First submitted 2019-02-28; First posted 2019-03-04 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Bowel Disease
Keywords: colonoscopy; biosignals; pain; sedation
MeSH Terms: conditions — Intestinal Diseases; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Nurse-administered propofol sedation has become the standard procedure for colonoscopy in Germany. Although patient satisfaction with this method is high, there is little data about the satisfaction of the examiner and factors that might negatively influence this satisfaction. Often due to the fact that the sedated patient usually expresses pain by movements of the body and paralinguistic sounds the examination has to pause until the next propofol bolus induces a deeper sedation. In order to measure the correlation of examiner satisfaction and negative factors the investigators initiated this prospective observational study. During this study examiner satisfaction and the correlation with observer reported pain (movements and paralinguistic sounds) will be measured. Additionally different biopotentials (electromyography, skin conductance level, body temperature, pulse) of the patient will be recorded during the examination and feature pattern will be correlated to the observer reported pain in order to detect pain before the expression of pain leads to a pause in the colonoscopy examination. Other factors that might influence examiner satisfaction, like duration to reach the caecum and duration of polypectomy will additionally be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18
* ASA classification I to II
* Indication for colonoscopy with propofol sedation
* Written informed consent

Exclusion Criteria:

* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled at the University Hospital for a colonoscopy using propofol sedation.
Sampling Method: Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Correlation between clinician satisfaction with sedation and pain experienced during colonoscopy | 1 day
  Correlation between Clinician Satisfaction with Sedation Instrument (CSSI) and observer reported pain (movements and paralinguistic sounds) during sedation
Prediction of observer reported pain by biopotential feature pattern | 1 day
  Prediction of observer reported pain events (movements and paralinguistic sounds) by biopotential feature pattern.

SECONDARY OUTCOMES:
Correlation between clinician satisfaction with sedation (CSSI) and sedation depth | 1 day
  Correlation between clinician satisfaction with sedation (CSSI) and sedation depth measured by Modified Observer's assessment of Alertness/Sedation Score
Correlation between clinician satisfaction with sedation (CSSI) and frequency of sedation use | 1 day
  Correlation between clinician satisfaction with sedation (CSSI) and frequency of sedation use measured in relation to total examination duration.
Correlation between clinician satisfaction with sedation (CSSI) and resected polyp count | 1 day
  Correlation between clinician satisfaction with sedation (CSSI) and resected polyp count
Correlation between clinician satisfaction with sedation (CSSI) and total polyp resection time | 1 day
  Correlation between clinician satisfaction with sedation (CSSI) and total polyp resection time
Correlation between clinician satisfaction with sedation (CSSI) and time to reach caecum | 1 day
  Correlation between clinician satisfaction with sedation (CSSI) and time to reach caecum
Correlation between clinician satisfaction with sedation (CSSI) and years of experience of assisting nurse | 1 day
  Correlation between clinician satisfaction with sedation (CSSI) and years of experience of assisting nurse

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Hann, Principal Investigator — University Ulm
Locations (1):
- University Ulm, Ulm, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hann A, Gruss S, Goetze S, Mehlhase N, Frisch S, Walter B, Walter S. Autonomous Nervous Response During Sedation in Colonoscopy and the Relationship With Clinician Satisfaction. Front Med (Lausanne). 2021 Jun 16;8:643158. doi: 10.3389/fmed.2021.643158. eCollection 2021. PMID 34222272